CLINICAL TRIAL: NCT06211101
Title: Evaluation of the Effectiveness of the Utilization of the Kangaroo Care Guide in the Neonatal Intensive Care Unit: An Evidence Utilization Study
Brief Title: Evaluation of the Effectiveness of the Utilization of the Kangaroo Care Guide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SelcukU-12-2023
Record Dates: First submitted 2023-12-21; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Kangaroo Care Trainig
Keywords: Kangaroo Care; trainig; Nurse; NICU

STUDY DESIGN:
Intervention Model Description: parallel group (experimental-control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Nurses were trained on the kangaroo care guide. Online training was given to neonatal nurses on the kangaroo care guide created by the researcher in line with the literature.
  Interventions: Other: Providing training on kangaroo care guide
- No Intervention: Control Group (No Intervention): Nurses weren't trained on the kangaroo care guide.

INTERVENTIONS:
Other: Providing training on kangaroo care guide — Online training was given to neonatal nurses on the kangaroo care guide created by the researcher in line with the literature.
  Arms: Experimental: Intervention Group

SUMMARY:
The aim of this study was to determine the effect of kangaroo care guideline-based training for nurses on nurses' knowledge level, kangaroo care practices and Attitude Towards Evidence-Based Nursing scale scores.

The study was parallel group (experimental-control), randomized controlled experimental design with pretest-posttest design.

It was carried out in the neonatal intensive care unit of Selçuk University Faculty of Medicine Hospital in Konya province. Study data were collected from 32 newborn nurses between October 2022 and January 2023. Premature infants in the intervention (n = 16) and control groups (n = 16) were determined by randomization method.

DETAILED DESCRIPTION:
Neonatal nurses in the intervention group were trained on the kangaroo care guide, but no application was made to the control group. Data were collected using the BP Information Form, BP Practice status, and the Attitudes Toward Evidence-Based Nursing Scale. Data were collected as a pretest before the application and as a posttest after the application. Pearson Chi-Square Test, Yates Correction and Fisher's Exact Test were used to compare categorical data according to groups. Two Independent Sample t Test was used to compare normally distributed variables and Mann Whitney U Test was used to compare non-normally distributed variables. Statistical significance level was accepted as p˂0.05.

ELIGIBILITY:
Inclusion Criteria:

* Having been working as a nurse in the Neonatal Intensive Care Unit for at least 6 months
* Volunteer

Exclusion Criteria:

* Working as a resuscitation nurse in the unit
* Being on maternity leave

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Kangaroo care information form | Change from baseline and post test (15 days later).
  It contains information questions about kangaroo care in line with the literature.
Kangaroo care application status | Change from baseline and post test (15 days later).
  It determines the application status of kangaroo care application steps.
Attitude Scale Towards Evidence-Based Nursing | Change from baseline and post test (15 days later).
  The scale consists of three subscales (Beliefs and expectations, Implementation intention and Emotions) and 15 items.
  The scale is a 5-point Likert type (1=strongly disagree, 2=disagree, 3=somewhat agree, 4=agree, 5=completely agree).
  The lowest score from the scale is 15 points and the highest score is 75 points. A high score indicates a positive attitude towards evidence-based nursing.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya, Selcuklu
  - Selcuk University, Konya

IPD SHARING:
Plan to Share IPD: No